CLINICAL TRIAL: NCT00647218
Title: A Pilot Study of Neoadjuvant Paclitaxel and Concurrent Radiation With Correlative Molecular Studies in Stage II/III Breast Cancer
Brief Title: Paclitaxel and Radiation Therapy in Treating Patients Undergoing Surgery for Stage II or Stage III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC BRE 9936; P30CA068485 (NIH); VU-VICC-BRE-9936
Record Dates: First submitted 2008-03-28; First posted 2008-03-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Post-operative adjuvant therapy; Drug: neoadjuvant therapy; Procedure: therapeutic surgical procedure; Radiation: Radiation therapy with concurrent Paclitaxel; Drug: Hormonal Therapy

INTERVENTIONS:
Drug: Post-operative adjuvant therapy — Adriamycin 60 mg/m2 IV over 20 minutes and Cytoxan 600 mg/m2 IV over 1 hour will be given every three weeks for 4 cycles.
  Other Names: None noted
Drug: neoadjuvant therapy — Paclitaxel 175 mg/m2 IV every 3 weeks x 3 cycles
  Other Names: None noted
Procedure: therapeutic surgical procedure — Modified radical mastectomy or segmental mastectomy plus axillary dissection 6-8 weeks following completion of chemotherapy/Radiotherapy.
  Other Names: None noted
Radiation: Radiation therapy with concurrent Paclitaxel — Radiation to breast 4680 cGy/26 fractions with concurrent Paclitaxel 30 mg/m2, twice per week
  Other Names: None noted
Drug: Hormonal Therapy — After completion of postoperative adjuvant Adriamycin and Cytoxan, hormonal therapy should be given at the discretion of the treating physician for all post-menopausal ER and/or PR positive patients. It is also recommended for pre-menopausal patients who are ER and/or PR positive.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving paclitaxel and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This clinical trial is studying how well giving paclitaxel together with radiation therapy works in treating patients undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of paclitaxel and concurrent radiotherapy (as measured by pathologic response rates) in patients with stage II or III breast cancer.

Secondary

* Evaluate the toxicities of this treatment regimen.
* Correlate paclitaxel-induced tumor response with local recurrence-free survival, distant disease-free survival, and overall survival.
* Evaluate protein expression profiles by mass spectrometry in biopsy material and blood specimens collected before and after treatment with paclitaxel.

OUTLINE:

* Neoadjuvant chemotherapy: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Chemoradiotherapy: Beginning 3-4 weeks after completion of neoadjuvant chemotherapy, patients receive paclitaxel IV over 1 hour twice weekly and undergo radiotherapy once daily, 5 days a week, for 6½ weeks.
* Surgery: At 6-8 weeks after completion of chemoradiotherapy, patients undergo surgical resection (e.g., modified radical mastectomy or lumpectomy and axillary node dissection).
* Adjuvant chemotherapy: Beginning 4-6 weeks after surgery, patients receive doxorubicin hydrochloride IV over 20 minutes and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Hormonal therapy: After completion of adjuvant chemotherapy, patients with estrogen receptor- and/or progesterone receptor-positive tumor receive hormonal therapy at the discretion of the treating physician.

Patients undergo blood and tissue sample collection periodically to analyze changes in cell cycle by flow cytometry; antibody assays; kinase assays for cyclin B1/CDC2; genetic assays for p53, p21, and other molecular markers; and protein expression assays by mass spectrometry.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically documented invasive carcinoma of the breast*

  * Tumor ≥ 2 cm in greatest dimension (e.g., T2-4) and any nodal status (e.g., N0-3), including locally advanced disease, as defined by the following criteria:

    * Primary tumor ≥ 5 cm
    * Tumor of any size with direct extension to the chest wall or skin
    * Inflammatory breast cancer (T4d)
    * Metastasis to ipsilateral internal mammary node
    * Ipsilateral lymph nodes that are clinically fixed to each other or to other structures (N2) NOTE: *Diagnosis may be made by core or tru-cut biopsies
* Measurable or evaluable tumor

  * Measurable disease is defined as any mass that can be reproducibly measured in two perpendicular dimensions
  * Evaluable disease is defined as any lesion visible by mammogram or palpable by physical exam that does not fit the above criteria of measurability
* Planning to undergo breast conservation surgery
* Willing to undergo AND is a candidate for radiotherapy, in the judgement of the treating radiation oncologist
* No evidence of distant metastatic disease (e.g., lung, liver, bone, brain)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Left ventricular ejection fraction ≥ 45%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancies within the past 5 years, except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No history of hypersensitivity reaction to products containing polysorbate 80 (Tween 80)
* No serious medical illness that, in the judgment of the treating physician, places the patient at risk
* No peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* Prior tamoxifen as chemoprevention allowed
* No prior radiotherapy to the ipsilateral breast

  * Prior radiotherapy to the contralateral breast is allowed
* No prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-02; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | 9 weeks

SECONDARY OUTCOMES:
Toxicity paclitaxel and radiation | at 18 weeks
Correlation of tumor response with local recurrence-free survival, distant disease-free survival, and overall survival | at time of disease progression or death by any cause
Protein expression profiles as measured by mass spectrometry before and after treatment with paclitaxel | Baseline and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Williamson Medical Center, Frankling, Tennessee
  - Jackson-Madison Hospital, Jackson, Tennessee
  - Boston Baskin Cancer Center, Memphis, Tennessee
  - Methodist Lebonheur Healthcare, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Cetner, Nashville, Tennessee